CLINICAL TRIAL: NCT07177001
Title: The Prevalence of Neck Pain and Low Back Pain in Physical Therapy Students at The University of the West Indies, Mona, Jamaica
Brief Title: Neck and Low Back Pain in Physical Therapy Students at The University of the West Indies, Mona, Jamaica
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Collaborators: The University of The West Indies, Mona (Unknown)
Responsible Party: Principal Investigator, Paula Dawson, MBBS, Head, Physical Medicine and Rehabilitation. Principal Investigator, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CREC-MN.0228,2024/2025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Back Pain; Low Back Pain; Musculoskeletal Pain; Spine Health; Physical Therapy; Physiotherapist Students; Physiotherapy; Rehabilitation; Neck Pain
Keywords: lower back pain; low back pain; neck pain; musculoskeletal pain; spine health; physical therapy students; physiotherapy students; rehabilitation
MeSH Terms: conditions — Back Pain; Low Back Pain; Musculoskeletal Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Control (Group A) (Experimental): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group A will be given a non-specific spine exercise program over an eight (8) week period after which time, participants will be reassessed using the CMDQ and NRS, as well as a Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain.
  Interventions: Behavioral: Clinical Control Group (Group A)
- Spine Exercise Program (Group B) (Experimental): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group B will be given a standardised spine-specific exercise program over an eight (8) week period, after which time they will be be reassessed using the CMDQ and NRS, as well as Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, having received the intervention.
  Interventions: Behavioral: Spine Exercise Program (Group B)

INTERVENTIONS:
Behavioral: Clinical Control Group (Group A) — The participants who reported the presence of neck or low back pain and were assigned to the clinical control group (Group A) after randomisation will receive a non-specific spine exercise program provided in a handout. The interventional group (Group B) will be asked to keep the standardised spine-specific exercise program confidential and not share with the control group (Group A). After eight (8) weeks, Group A participants will receive: the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess for changes in the frequency, discomfort and interference with work due to musculoskeletal pain; a Questionnaire B, to ascertain any changes in their pain level using the Numeric Rating Scale (NRS); as well as their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain.
  Arms: Clinical Control (Group A)
Behavioral: Spine Exercise Program (Group B) — The standardised spine-specific exercise program will be provided in a handout and given only to the intervention group (Group B), and will include specific spine basic neck or low back exercises to be done three (3) times per week, as well as brief stretching exercises, to be done during periods of sitting for greater than sixty (60) minutes. The selected participants will be asked to comply with instructions on the handout. Participants who experience worsening of their symptoms, or who develop new symptoms will be assessed as having an adverse outcome and will be withdrawn from the study and referred for evaluation and treatment if necessary.
  Arms: Spine Exercise Program (Group B)

SUMMARY:
The purpose of this study is to identify the prevalence of neck and low back pain in physical therapy students enrolled at the University of the West Indies, Mona; to assess their knowledge, attitude and practice of good spine health and to determine the outcome of a standardised spine exercise program on physical therapy students experiencing neck and low back pain, using a prospective randomised control design.

DETAILED DESCRIPTION:
Neck and low back pain are common musculoskeletal problems that affect most persons at some point in their lives, cutting across various professions. These conditions may be self-limiting, but in many cases, they become disabling and significantly impact productivity, social life, and activities of daily living. It is estimated that approximately 37% of back pain is associated with occupational factors. Prolonged sitting and awkward postures considerably increase the risk of low back pain, while neck pain is closely linked to slouching and repeated or prolonged neck movements. Health care professionals, including physical therapists, are one such group highly susceptible to musculoskeletal pain, and this vulnerability begins as early as their training years. Physical therapy training involves both preclinical and clinical phases that expose students to unique risk factors. During the preclinical period of training, physiotherapy students spend long hours sitting during lectures, studying, and completing assignments, often with sustained use of computers or electronic devices. In the clinical periods, students are immersed in a physically demanding training environment involving prolonged standing, manual patient handling and therapeutic exercises. A systematic review by Smith et al. found that low back pain was reported by 60-80% of physical therapy students during their education. Similarly, Johnson et al. revealed that 66.8% of physical therapy students experienced low back pain, with a significant proportion reporting limitations in daily activity. Comparative studies suggest that physical therapy students are at even higher risk of low back pain than medical students, with prevalence rates of 77.9% versus 54.3%, respectively. This difference is attributed to the physical nature of physical therapy training, which requires manual therapy techniques, patient transfers, and prolonged standing during clinical practice. Neck pain is also highly prevalent among physical therapy students. Brown et al. reported a 69% prevalence of neck pain among physical therapy undergraduate students, most of whom attributed symptoms to prolonged studying, poor posture, and excessive electronic device use. Regional studies in Saudi Arabia and Pakistan further reported neck pain prevalence rates of 48.8% and 51.8%, respectively, with postural strain, poor ergonomics, and psychosocial stress identified as major contributors. Risk factors for neck and low back pain pain among physical therapy students are therefore multifactorial, including poor ergonomics while studying or performing manual techniques, the physical demands of training such as lifting patients and prolonged standing, sedentary behaviours during study periods, and psychosocial stress arising from academic pressure. Although physical therapy students are trained in exercise science, their personal levels of physical activity may vary, which may further influence susceptibility to musculoskeletal pain. Exercise therapy is one of the most effective non-pharmacological interventions for musculoskeletal pain. Chou and Huffman (2007), in their review of non-pharmacologic therapies for acute and chronic low back pain, demonstrated significant improvements in both pain reduction and function with exercise compared to other interventions. Exercise enhances spinal strength, flexibility, and stability, while promoting nutrient transfer to discs, ligaments, and soft tissues, thereby reducing the likelihood of injury. Low back and core-strengthening exercises, in particular, are widely regarded as an optimal approach to restoring spinal balance and alleviating pain.

At the University of the West Indies (UWI), Mona, there are currently 120 physical therapy students enrolled across three years, with approximately 40 students per cohort. This study seeks to determine the prevalence of neck and low back pain in physical therapy students, to assess their knowledge, attitude, and practice regarding spine health, and to evaluate the outcome of a standardised spine-specific exercise program on reducing pain and improving functional status. Students reporting pain will be prospectively randomised into control and intervention arms, with the latter receiving the standardised spine-specific exercise program over an eight (8) weeks period. Outcome measures will include the Numeric Rating Scale (NRS), the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ), and structured questionnaires to assess function, knowledge, attitude, and practice. To the best of the researcher's knowledge, this will be the first randomised controlled study conducted in the Caribbean investigating the prevalence of neck and low back pain among physical therapy students, while simultaneously assessing the effectiveness of a targeted exercise based intervention.

ELIGIBILITY:
Inclusion Criteria:

1. All students enrolled in the Physical Therapy program at the University of the West Indies, Mona Campus, Jamaica during the period November 1, 2025 to October 31, 2026.
2. Individuals who express a willingness to consent to the study.
3. Individuals who express a willingness to adhere to the standardised exercise program for the stipulated period.

Exclusion Criteria:

1. Individuals with a history of having spine surgery.
2. Individuals who were previously diagnosed with spine pathology and currently receiving rehabilitation therapy.
3. Individuals who express an unwillingness to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender men and cisgender women
Enrollment: 120 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | From enrollment to the end of treatment at eight (8) weeks
  The Cornell Musculoskeletal Discomfort Questionnaire measures the frequency, discomfort and interference with work due to musculoskeletal pain, as reported by participants. The individually reported frequency score is then multiplied by the discomfort score and by the interference score to determine overall severity of pain experienced. This tallied score is then classified by severity into: no discomfort (0), mild (1 to 4.5), moderate (5 to 14), severe (15 - 45) and very severe (45 or higher). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their reported scores.

SECONDARY OUTCOMES:
Knowledge, Attitude and Practice towards Musculoskeletal Problems of Neck and Low back Pain (Questionnaire A) | Done at the time of enrollment (Baseline)
  Questionnaire A is a self-administered general questionnaire used to evaluate knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in Knowledge, Attitude and Practice Towards Musculoskeletal Problems of Neck and Low Back Pain (Questionnaire B) | From Enrollment to the end of treatment at 8 weeks
  Questionnaire B is a self-administered general questionnaire used to evaluate changes in knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in the Numeric Rating Scale (NRS) | From Enrollment to the end of treatment at 8 weeks
  The Numeric Rating Scale is a reliable and valid, unidimensional 11-point scale used for patient self-reporting of perceived pain. Its scale uses integers which range from zero (0) to ten (10), where 0 represents no pain, and 10 represents the worst imaginable pain. This is then categorised into mild (1-3), moderate (4-6), and severe (7-10). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their perceived pain. This scale is from public domains and as such, permission for its use is not required.

CONTACTS AND LOCATIONS:
Overall Officials: Paula U.A Dawson, MBBS, Diplomate ABPMR, Principal Investigator — Division of Physical Medicine and Rehabilitation, Faculty of Medical Sciences, The University of the West Indies, Mona, Jamaica.
Locations (1):
- Faculty of Medical Sciences Teaching and Research Complex, University of The West Indies-Mona Campus, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogunlana MO, Govender P, Oyewole OO. Prevalence and patterns of musculoskeletal pain among undergraduate students of occupational therapy and physiotherapy in a South African university. Hong Kong Physiother J. 2021 Jun;41(1):35-43. doi: 10.1142/S1013702521500037. Epub 2021 Jan 18. PMID 34054255
- [Background] Naing L, Nordin RB, Abdul Rahman H, Naing YT. Sample size calculation for prevalence studies using Scalex and ScalaR calculators. BMC Med Res Methodol. 2022 Jul 30;22(1):209. doi: 10.1186/s12874-022-01694-7. PMID 35907796
- [Background] Erdinc O, Hot K, Ozkaya M. Turkish version of the Cornell Musculoskeletal Discomfort Questionnaire: cross-cultural adaptation and validation. Work. 2011;39(3):251-60. doi: 10.3233/WOR-2011-1173. PMID 21709361
- [Background] Ariens GA, van Mechelen W, Bongers PM, Bouter LM, van der Wal G. Physical risk factors for neck pain. Scand J Work Environ Health. 2000 Feb;26(1):7-19. doi: 10.5271/sjweh.504. PMID 10744172
- [Background] Standaert CJ, Herring SA. Expert opinion and controversies in musculoskeletal and sports medicine: core stabilization as a treatment for low back pain. Arch Phys Med Rehabil. 2007 Dec;88(12):1734-6. doi: 10.1016/j.apmr.2007.10.002. PMID 18047895
- [Background] Gordon R, Bloxham S. A Systematic Review of the Effects of Exercise and Physical Activity on Non-Specific Chronic Low Back Pain. Healthcare (Basel). 2016 Apr 25;4(2):22. doi: 10.3390/healthcare4020022. PMID 27417610
- [Background] O'Sullivan PB, Phyty GD, Twomey LT, Allison GT. Evaluation of specific stabilizing exercise in the treatment of chronic low back pain with radiologic diagnosis of spondylolysis or spondylolisthesis. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2959-67. doi: 10.1097/00007632-199712150-00020. PMID 9431633
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] Garcia L, Thompson J, Reed B. Low back pain in nursing students: Prevalence and risk factors. Nurs Educ Perspect. 2019;35(3):150-156.
- [Background] Williams N, Garcia M, Robinson P. Musculoskeletal pain in healthcare students: A comparative analysis. J Allied Health Sci. 2021;37(4):210-222.
- [Background] Khan F, Tariq H, Malik Z. The impact of poor posture on neck pain among undergraduate physiotherapy students. Pak J Rehabil. 2021;10(1):78-85.
- [Background] Ali S, Hassan R, Ahmed M. Prevalence of neck among physiotherapy students in Saudi Arabia. Saudi J Health Sci. 2020;9(2):45-51.
- [Background] Brown P, Clark M, Adams T. Neck pain prevalence and associated risk factors among physiotherapy students. J Musculoskeletal Pain 2022;29(3):183-194.
- [Background] Doe J, Smith L, Wilson H. Comparison of musculoskeletal disorders in physiotherapy and medical students. J Med Educ Res. 2019;40(2):115-124.
- [Background] Johnson D, Miller K, Lee R. Low back pain among physiotherapy students: A cross sectional study. Physiother Res Int. 2021;28(1):e1872.
- [Background] Smith A, Jones B, Patel C. The prevalence and impact of low back pain in physiotherapy students: A systematic review. J Rhys There Sci 2020;32(4):567-574.
- [Background] Smith DR, Leggat PA, Walsh LJ. Workplace hazards among Australian dental students. Aust Dent J. 2009 Jun;54(2):186-8. doi: 10.1111/j.1834-7819.2009.01116_8.x. No abstract available. PMID 19473172
- [Background] Lorusso A, Vimercati L, L'abbate N. Musculoskeletal complaints among Italian X-ray technology students: a cross-sectional questionnaire survey. BMC Res Notes. 2010 Apr 24;3:114. doi: 10.1186/1756-0500-3-114. PMID 20416101
- [Background] Smith DR, Leggat PA. Musculoskeletal disorders among rural Australian nursing students. Aust J Rural Health. 2004 Dec;12(6):241-5. doi: 10.1111/j.1440-1854.2004.00620.x. PMID 15615575
- [Background] Alshagga MA, Nimer AR, Yan LP, Ibrahim IA, Al-Ghamdi SS, Radman Al-Dubai SA. Prevalence and factors associated with neck, shoulder and low back pains among medical students in a Malaysian Medical College. BMC Res Notes. 2013 Jul 1;6:244. doi: 10.1186/1756-0500-6-244. PMID 23815853
- [Background] Falavigna A, Teles AR, Mazzocchin T, de Braga GL, Kleber FD, Barreto F, Santin JT, Barazzetti D, Lazzaretti L, Steiner B, Beckenkamp NL. Increased prevalence of low back pain among physiotherapy students compared to medical students. Eur Spine J. 2011 Mar;20(3):500-5. doi: 10.1007/s00586-010-1646-9. Epub 2010 Dec 7. PMID 21136121
- [Background] Smith DR, Wei N, Ishitake T, Wang RS. Musculoskeletal disorders among Chinese medical students. Kurume Med J. 2005;52(4):139-46. doi: 10.2739/kurumemedj.52.139. PMID 16639985
- [Background] Lis AM, Black KM, Korn H, Nordin M. Association between sitting and occupational LBP. Eur Spine J. 2007 Feb;16(2):283-98. doi: 10.1007/s00586-006-0143-7. Epub 2006 May 31. PMID 16736200
- [Background] Punnett L, Pruss-Utun A, Nelson DI, Fingerhut MA, Leigh J, Tak S, Phillips S. Estimating the global burden of low back pain attributable to combined occupational exposures. Am J Ind Med. 2005 Dec;48(6):459-69. doi: 10.1002/ajim.20232. PMID 16299708
- [Background] Ehrlich GE. Low back pain. Bull World Health Organ. 2003;81(9):671-6. Epub 2003 Nov 14. PMID 14710509